CLINICAL TRIAL: NCT06183554
Title: CXCR4 Targeted PET Imaging in the Diagnosis and Identification of Primary Aldosteronism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiao Chen (Other)
Responsible Party: Sponsor-Investigator, Xiao Chen, Director of Nuclear Medicine Department, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Other Study IDs: 2023239
Record Dates: First submitted 2023-12-14; First posted 2023-12-27 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Primary Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — adrenal resection specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CXCR4 — Patients with clinical suspected primary aldosteronism will receive a CXCR4 PET imaging.

SUMMARY:
This study aimed to prospectively evaluate the utility of C-X-C chemokine receptor type 4 (CXCR4) positron emission tomography (PET) imaging in patients with clinical suspected primary aldosteronism (PA), with postoperative pathological or follow-up results as reference standards.

DETAILED DESCRIPTION:
1. Record the course of disease, the laboratory examination (e.g., potassium, aldosterone, aldosterone-to-renin ratio, intravenous salt-loading test or captopril test) and the results of adrenal vein sampling in patients with clinically suspected PA.
2. PET image analysis: Record and evaluate the following indicators: the maximum standardized uptake value (SUVmax) of lesions, the mean standardized uptake value (SUVmean) of normal liver, the SUVmean of adjacent normal adrenal tissue, the ratio of the lesional SUVmax to the normal liver SUVmean (LLR), and the ratio of the lesional SUVmax to the adjacent adrenal tissue SUVmean (LAR).
3. Pathological analysis: Hematoxylin and eosin staining and immunohistochemical analyses will be performed. Immunohistochemical analysis will be used to investigate the expression of aldosterone synthase (CYP11B2) and CXCR4.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent hypertension with blood pressure > 150/100 mmHg, refractory hypertension (blood pressure >140/90 mmHg with combined use of three types of antihypertensive medications, including diuretics), or with hypokalemia of blood pressure >140/90 mmHg;
2. Refractory hypertension with an aldosterone-to-renin ratio (ARR) ≥ 2.0 (ng/dl)/(mU/L);
3. Positive intravenous salt-loading test or captopril test;
4. Hypertension and adrenal lesions;
5. Patient ≥18 years of age at the time of consent;
6. Provided written informed consent authorisation before participating in the study.

Exclusion Criteria:

1. Refusal by the patients to undergo CXCR4 PET imaging, adrenal vein sampling, superselective adrenal arterial embolization or adrenalectomy;
2. Suspicion of familial hyperaldosteronism type 1 (FH-1) or type 3 (FH-3)；
3. Suspicion of adrenocortical carcinoma；
4. Severe comorbidity potentially interfering with treatment or HRQoL；
5. Requirement of medication interfering with the study protocol；
6. Pregnancy or lactation；
7. Estimated glomerular filtration rate <40 mL/min/1.73 m².

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects the investigators selected are adults who are not restricted by gender.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Standardised uptake values | completed within one week after the PET examination
  Standardised uptake values of suspected adrenal disease in CXCR4 PET imaging

SECONDARY OUTCOMES:
Immunohistochemical results | completed within one week after surgery
  Immunohistochemical evaluation of postoperative adrenal specimens

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Chen, Ph.D, Principal Investigator — Daping Hospital, Army Medical University
Locations (1):
- Department of Nuclear Medicine, Daping Hospital of Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu J, Xu T, Shen H, Song Y, Yang J, Zhang A, Ding H, Xing N, Li Z, Qiu L, Ma L, Yang Y, Feng Z, Du Z, He W, Sun Y, Cai J, Li Q, Chen Y, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Accuracy of Gallium-68 Pentixafor Positron Emission Tomography-Computed Tomography for Subtyping Diagnosis of Primary Aldosteronism. JAMA Netw Open. 2023 Feb 1;6(2):e2255609. doi: 10.1001/jamanetworkopen.2022.55609. PMID 36795418